CLINICAL TRIAL: NCT04412473
Title: COVID-19 Respiratory Distress and Antithrombotic Drugs inSubject's Habits
Brief Title: COVID-19 Respiratory Distress and Antithrombotic Drugs in Subject's Habits
Acronym: CRASH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7837
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2
Keywords: Sars-CoV2; Covid-19; Antithrombotic treatments; ARDS; Hypoxemia; Thrombosis; Pulmonary arteries; Endothelial
MeSH Terms: conditions — COVID-19; Hypoxia; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current management of VID-19 consists of oxygen support without specific treatment. Hospitalization may suddenly require delayed resuscitation. This evolution corresponds to an atypical acute respiratory distress syndrome (ARDS), the mechanism of which is poorly understood and difficult to predict. The general pathophysiology of ARDS, the vascular tropism of SARS-Cov2, the description of coagulopathy and numerous pulmonary artery thromboses in resuscitation and the encouraging investigation of antithrombotics in general ARDS

ELIGIBILITY:
Inclusion Criteria:

* Major Subject (≥18 years)
* Subject hospitalised in HUS or GHRMSA for COVID-19
* The diagnosis COVID-19 confirmed by smear or evoked by CT scan or chest X-ray without a differential diagnosis retained in the medical record
* Subjects who, after being informed, do not wish to have their data reused for the purposes of this research

Exclusion Criteria:

* Subject who expressed opposition to participating in the study
* Subject under guardianship or trusteeship
* Subject under safeguard of justice
* Patient hospitalized in a geriatric service or in a ward not labeled COVID (surgery, oncology,...) or in a short-term hospitalization unit without transfer to another service.
* Serious patient on admission to the emergency room and recused from resuscitation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult Partients hospitalised in HUS or GHRMSA for COVID-19 with diagnosis COVID-19 confirmed by smear or evoked by CT scan or chest X-ray without a differential diagnosis retained in the medical record
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Analysis of Respiratory Distress and Antithrombolytic Therapy in Patients with covid19 | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service Médecine Intensive et Réanimation, Strasbourg, France